CLINICAL TRIAL: NCT01194401
Title: A Prospective, Non-interventional Multi-center Observational Study to Evaluate the Long-term Effectiveness and Safety of Tocilizumab in Patients With Active Rheumatoid Arthritis in Daily Practice
Brief Title: An Observational Study on Long-Term Effectiveness and Safety of RoActemra/Actemra (Tocilizumab) in Daily Practice in Patients With Rheumatoid Arthritis (ICHIBAN)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22928
Record Dates: First submitted 2010-09-01; First posted 2010-09-03 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This prospective, multi-center observational study will assess the long-term efficacy and safety of RoActemra/Actemra in daily practice in patients with active moderate to severe rheumatoid arthritis who have an inadequate response or are intolerant to one or more disease-modifying antirheumatic drugs (DMARDs) or tumour necrosis factor (TNF) antagonists. Data will be collected from patients initiated on RoActemra/Actemra treatment according to label by decision of the treating physician. Anticipated time for data collection from each patient will be 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Active moderate to severe rheumatoid arthritis
* Inadequate response or intolerant to previous therapy with one or more disease-modifying antirheumatic drugs (DMARDs) or tumour necrosis factor (TNF) antagonists
* Prescription of RoActemra/Actemra according to label

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with inadequate response or intolerant to DMARDs and anti-TNF
Sampling Method: Probability Sample
Enrollment: 3404 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with clinical remission defined as disease activity score DAS28 < 2.6 | 5 years

SECONDARY OUTCOMES:
Time to DAS28 remission | 5 years
Proportion of patients with good or moderate response according to EULAR criteria | 5 years
Time to good or moderate response according to EULAR criteria | 5 years
Factors related to response (C-reactive protein, rheumatoid factor, inadequate response to DMARDs or anti-TNF, duration of illness) | 5 years
Dose-modifications and discontinuations of RoActemra/Actemra | 5 years
Safety: Incidence of adverse events | 5 years
Efficacy of other possible RA therapies in case of inadequate response to RoActemra/Actemra (DAS28, EULAR criteria) | 5 years
Safety of other possible RA therapies in case of inadequate response to RoActemra/Actemra (adverse events) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Osnabrück, Germany